CLINICAL TRIAL: NCT07304076
Title: Clinical Research on the Comparative Effectiveness and Safety of JHG002 Therapy for Chronic Low Back Pain: A Multicenter Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2024-03
Record Dates: First submitted 2025-12-11; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: chronic low back pain; pharmacopuncture
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: 2-arm parallel multicenter RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hominis placental pharmacopuncture (Experimental): Participants in the experimental group will receive JHG002 pharmacopuncture twice weekly for 5 weeks (total 10 sessions). JHG002 (0.05-0.1 mL per point) will be administered to 8-10 acupuncture points commonly used for chronic low back pain, including BL23, BL24, BL25, GV3, and GV4, with optional GB30 based on symptoms.
  Interventions: Drug: Hominis placental pharmacopuncture
- Physical Therapy Group (Active Comparator): Participants in the control group will receive standardized transcutaneous electrical nerve stimulation (TENS) therapy twice weekly for 5 weeks (total 10 sessions). Each session will last 15 minutes and will be administered using a unified protocol across all participating sites to target the lumbar region.
  Interventions: Device: Tanscutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Drug: Hominis placental pharmacopuncture — JHG002 pharmacopuncture is a purified Hominis placenta extract formulated for injection at acupuncture points. In Korean medicine, Hominis placenta has traditionally been used to support vitality, relieve chronic pain, and enhance functional recovery.
  Other Names: JHG002
  Arms: Hominis placental pharmacopuncture
Device: Tanscutaneous electrical nerve stimulation (TENS) — Transcutaneous electrical nerve stimulation is a non-invasive physical therapy that delivers low-intensity electrical stimulation to the lumbar area to reduce pain and muscle tension.
  Other Names: TENS; electrical nerve stimulation
  Arms: Physical Therapy Group

SUMMARY:
A multicenter randomized controlled trial

DETAILED DESCRIPTION:
This multicenter, randomized, parallel-group controlled trial aims to evaluate the effectiveness and safety of JHG002 pharmacopuncture in adults with chronic low back pain lasting more than 6 months. A total of 96 participants will be randomly assigned in a 1:1 ratio to receive either JHG002 pharmacopuncture or standard physical therapy with transcutaneous electrical nerve stimulation (TENS).

Participants in the JHG002 group will receive 10 treatment sessions over 5 weeks (twice weekly), with 0.05-0.1 mL of JHG002 administered to 8-10 acupuncture points commonly used for lumbar pain. The control group will receive standardized TENS therapy twice weekly for 15 minutes per session during the same treatment period.

Outcome assessments will be conducted at baseline and Weeks 1, 2-5, 9, 6, 13, and 25. The primary outcome is the change in low back pain intensity measured by the Numeric Rating Scale (NRS) at Week 6. Secondary outcomes include radiating leg pain NRS, visual analogue scale (VAS) scores, functional disability (Oswestry Disability Index; 6-item Roland-Morris Disability Questionnaire), quality of life (EQ-5D-5L; HINT-8), patient global impression of change (PGIC), credibility/expectancy, analgesic use, and economic outcomes such as direct/indirect medical costs and productivity loss.

Safety will be assessed through adverse event monitoring, vital signs, laboratory tests, and concomitant medication review. Adverse events will be evaluated according to WHO-UMC causality and standard severity grading. The study will follow a 4-year timeline from IRB approval to final follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 to 69 years at the time of signing the informed consent.
* Individuals who have experienced low back pain for ≥6 months, presenting with either continuous or intermittent symptoms.
* Participants with a Numeric Rating Scale (NRS) score ≥ 5 for low back pain at screening.
* Individuals who fully understand the clinical trial procedures and voluntarily agree to participate by providing written informed consent.

Exclusion Criteria:

* Patients diagnosed with serious underlying conditions that may cause low back pain, such as spinal metastasis of malignancy, acute vertebral fracture, or spinal dislocation.
* Patients with progressive neurological deficits or those presenting with severe neurological symptoms.
* Patients whose pain originates from non-spinal soft tissue disorders, including tumors, fibromyalgia, rheumatoid arthritis, or gout.
* Individuals with other chronic medical conditions that may interfere with treatment response or interpretation of study outcomes, such as stroke, myocardial infarction, chronic kidney disease, diabetic neuropathy, dementia, or epilepsy.
* Individuals currently taking corticosteroids, immunosuppressants, psychiatric medications, or any other drugs that may influence study results.*
* Patients for whom pharmacopuncture is inappropriate or unsafe, including those with bleeding disorders or those receiving anticoagulant therapy.
* Individuals who have taken analgesic medications such as NSAIDs or received pharmacopuncture treatment within the past 1 week.
* Women of childbearing potential who are unwilling to use medically acceptable contraception (e.g., surgical sterilization, intrauterine device, condom or diaphragm use, injectable or implantable contraceptives) throughout the study period.
* Pregnant or breastfeeding women.
* Individuals with a history of hypersensitivity or allergic reactions to Hominis placenta pharmacopuncture (JHG002).
* Patients with uncontrolled diabetes mellitus (fasting blood glucose ≥ 180 mg/dL).
* Individuals whose AST (GOT) or ALT (GPT) levels are ≥ 2 times the upper limit of the normal range at the study site.
* Individuals whose serum creatinine levels are ≥ 2 times the upper limit of the normal range at the study site.
* Patients suspected of having an underlying organic disease.
* Patients with moderate systemic complications involving organs other than the heart, liver, or kidneys.
* Patients with psychogenic disorders.
* Individuals with an implanted cardiac pacemaker.
* Patients with inflammation, infection, wounds, or other lesions at the planned pharmacopuncture sites that would prevent safe administration.
* Patients within 3 months after lumbar spine surgery.
* Individuals who have participated in another clinical trial within the past 1 month, or who plan to participate in another clinical trial-including follow-up periods-within 6 months from the screening date.
* Any individual deemed unsuitable for participation in this study by the investigator.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-12-17 (Estimated); Primary Completion 2029-11-28 (Estimated); Study Completion 2029-11-28 (Estimated)

PRIMARY OUTCOMES:
Change in low back pain intensity (NRS) | Week 1, 2-5, 6, 9, 13, 25
  The primary outcome is the change in low back pain intensity between baseline and Week 6. Low back pain severity during the past week will be assessed using the Numeric Rating Scale (NRS), where patients rate their pain on an 11-point scale ranging from 0 (no pain) to 10 (the worst pain imaginable). Participants will be instructed to report their average low back pain intensity over the past 7 days.

SECONDARY OUTCOMES:
Change in radiating leg pain intensity (NRS) | Week 1, 2-5, 6, 9, 13, 25
  Radiating leg pain severity will be evaluated using the same 0-10 Numeric Rating Scale (NRS), assessing the degree of pain or discomfort radiating from the lumbar region to the lower extremities. Participants will indicate the level of radiating pain they experienced during the past week, with higher scores representing greater severity.
Low back pain Visual Analogue Scale (VAS) | Week 1, 2-5, 6, 9, 13, 25
  The 100-mm Visual Analogue Scale (VAS) will be used to assess the intensity of low back pain. Participants will mark a point on a horizontal line anchored by "no pain" at the left end and "the most severe pain imaginable" at the right end. The distance in millimeters from the left end will be recorded as the pain score. This measure will be collected repeatedly to monitor pain trajectory over time.
Radiating leg pain Visual Analogue Scale (VAS) | Week 1, 2-5, 6, 9, 13, 25
  A VAS will also be used to evaluate radiating leg pain. Participants will indicate their perceived leg pain intensity on a 100-mm line in the same format used for the low back pain VAS. This measure provides a continuous index of radiating pain severity.
Oswestry Disability Index (ODI) | Weeks 1, 6, 13, 25
  The Oswestry Disability Index is a validated questionnaire assessing disability related to chronic low back pain. It consists of 10 items covering domains such as pain intensity, lifting, sitting, standing, sleep, and social life. Each item is scored from 0 to 5, and the total score is converted into a percentage (0-100%), with higher scores indicating greater functional impairment.
6-item Roland-Morris Disability Questionnaire (RMDQ-6) | Weeks 1, 6, 13, 25
  The RMDQ-6 is a short form of the Roland-Morris Disability Questionnaire that evaluates functional limitations in daily activities due to low back pain. The questionnaire consists of 6 binary (yes/no) items, and the total score ranges from 0 to 6. Higher scores reflect more severe disability.
Patient Global Impression of Change (PGIC) | Week 6, 13, 25
  PGIC is a single-item global assessment that measures the participant's overall perception of improvement or worsening after treatment. It uses a 7-point Likert scale, ranging from "very much improved" to "very much worse." This outcome captures the participant's subjective treatment benefit.
Health-related Quality of Life (EQ-5D-5L) | Weeks 1, 6, 13, 25
  The EQ-5D-5L evaluates quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each item has five response levels (no problems to extreme problems). The questionnaire also includes a 0-100 visual analogue scale to assess the participant's self-rated health status. Higher index values and VAS scores indicate better quality of life.
HINT-8 (Health-related Quality of Life Instrument) | Weeks 1, 6, 13, 25
  HINT-8 is a Korean-developed quality-of-life measurement tool consisting of eight items assessing physical, social, and mental health. Each item uses a 4-level response scale, and lower scores indicate better health status. This instrument is widely used in Korean health-economic studies.
Analgesic consumption | Week 1, 2-5, 6, 9, 13, 25
  Participants will record all use of rescue analgesic medications throughout the study period. Data will include type, dose, frequency, and duration of use. Increased analgesic intake may indicate worsening symptoms or insufficient treatment response.
Credibility and Expectancy Questionnaire | Screening
  This scale evaluates the participant's belief in the credibility and potential effectiveness of the assigned treatment. It includes both cognitive credibility items and emotional expectancy items, scored on Likert scales. Higher scores indicate greater perceived treatment plausibility and expected benefit.
Work Productivity and Activity Impairment Questionnaire (WPAI) | Week 1, 2-5, 6, 9, 13, 25
  The WPAI assesses the impact of low back pain on work performance and daily activities. It includes four domains: absenteeism, presenteeism, overall work impairment, and activity limitations. Scores are expressed as percentages, with higher percentages reflecting greater impairment.
Economic evaluation variables | Week 2
  Costs related to medical care, transportation, time burden, lost productivity, and indirect cost components will be collected to evaluate the cost-effectiveness of JHG002 compared with TENS. Data will be used for both cost-effectiveness and cost-utility analyses.

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Kyung Hee University Korean Medicine Hospital at Gangdong, Seoul, Gangdong-gu
  - Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, GGyeonggi-do
  - Dongguk University Bundang Oriental Hospital, Seongnam, GGyeonggi-do

IPD SHARING:
Plan to Share IPD: No